CLINICAL TRIAL: NCT02966080
Title: Fixed Low-dose Heparin Versus Standard Adjusted-dose Heparin Infusion in Adults Receiving Venovenous Extracorporeal Membrane Oxygenation (ECMO) With a Heparin Bonded Circuit.
Brief Title: Fixed Low-dose Heparin Versus Standard Adjusted-dose Heparin Infusion in Adults Receiving Venovenous ECMO With a Heparin Bonded Circuit.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled, study will not be conducted.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Robert Raschke, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1609884386
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Acute Respiratory Failure; Extracorporeal Membrane Oxygenation Complication; Bleeding
Keywords: extracorporeal membrane oxygenation; intravenous heparin
MeSH Terms: conditions — Hemorrhage | interventions — 1,7-dioxa-2,6-diaza-4,4-dioxide-4,7a-dithia-3H,5H-benzo(cd)pentalene; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjusted-dose heparin (Other): Patients in this arm of the study will receive intravenous unfractionated heparin at a dose adjusted to achieve an activated clotting time of 180-200 seconds.
  Interventions: Drug: HEP-IV
- Fixed low-dose heparin (Other): Patients in this arm of the study will receive intravenous unfractionated heparin at 500 units/hour without activated clotting time monitoring.
  Interventions: Drug: HEP-IV

INTERVENTIONS:
Drug: HEP-IV
  Other Names: heparin

SUMMARY:
Heparin is a blood thinner used to prevent blood clots in patients on a form of life-support called ECMO. Heparin can cause bleeding - the most common complication of ECMO. New materials used in ECMO machines may help prevent clots - this could allow the use of lower doses of heparin which might reduce the risk of bleeding. Our study will compare low dose to high dose heparin in patients on ECMO. We think low dose heparin may be adequate to prevent clotting, but may cause less bleeding and be safer for patients.

DETAILED DESCRIPTION:
Intravenous heparin is considered standard therapy to prevent clotting complications in patients on ECMO, however the optimal method of heparin dosing has not yet been determined. International surveys have shown that most ECMO centers use adjusted dose heparin to achieve an activated clotting time of at least 180 seconds. However, heparin may contribute to the most common complication of ECMO - bleeding. Advances in material technology have potentially reduced the thrombogenicity of modern ECMO circuits. Our observational data suggest that fixed low dose heparin infusion may reduce the rate of bleeding complications from 75% to 50% compared to standard adjusted-dose heparin, without increasing clotting complications. We intend to perform a randomized controlled trial in adults receiving venovenous ECMO comparing these two heparin regimens. The main outcome measures are bleeding complications and oxygenator failure due to clotting. A safety committee will monitor the results of the study. Power calculations indicate a sample size of 110 patients is required, which we estimate will take us five years to achieve.

ELIGIBILITY:
Inclusion Criteria:

* on ECMO for acute respiratory failure, achieving ECMO blood flow rate >3L/min,
* patient or surrogate able to speak/understand English or Spanish

Exclusion Criteria:

* History of heparin-induced thrombocytopenia, decision by clinicians to run ECMO off heparin due to high bleeding risk,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
significant bleeding complications | intraoperative
  requires surgery, >1 unit packed blood cell transfusion or is intracranial, pulmonary or retroperitoneal

SECONDARY OUTCOMES:
Oxygenator failure | intraoperative
  Requirement to replace oxygenator due to clotting
cerebral vascular event (stroke) | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Robert Raschke, MD, Principal Investigator — Banner University Medical Center
Locations (1):
- Banner - University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esper SA, Levy JH, Waters JH, Welsby IJ. Extracorporeal membrane oxygenation in the adult: a review of anticoagulation monitoring and transfusion. Anesth Analg. 2014 Apr;118(4):731-43. doi: 10.1213/ANE.0000000000000115. PMID 24651227
- [Background] Poulos EM, Raschke R, Amabile O et al. A Nonrandomized comparison of three different heparin infusion strategies for patients receiving venovenous extracorporeal membrane oxygenation. Am J Respir Crit Care Med 2014;189: A4499.
- See also: ELSO anticoagulation guideline — http://www.elso.org